CLINICAL TRIAL: NCT05160740
Title: Multicenter Randomized Controlled Clinical Trial of Indocyanine Green Molecular Fluorescence Imaging in the Diagnosis and Treatment of Primary Liver Cancer
Brief Title: Indocyanine Green Molecular Fluorescence Imaging Technique Using in Diagnosis and Treatment of Primary Liver Cancer
Acronym: ICGMFITinPLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Chihua Fang,MD, Clinical Professor, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-090-01
Record Dates: First submitted 2021-11-09; First posted 2021-12-16 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Liver Cancer
Keywords: indocyanine green; local resection
MeSH Terms: conditions — Liver Neoplasms | interventions — Indocyanine Green; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG molecular fluorescence imaging guided surgery (Experimental): ICG molecular fluorescence imaging will be used in local hepatectomy of primary liver cancer in this group
  Interventions: Drug: Indocyanine green for injection
- No ICG molecular fluorescence imaging guided surgery (Placebo Comparator): ICG molecular fluorescence imaging will not be used in local hepatectomy of primary liver cancer in this group
  Interventions: Drug: Indocyanine green for injection

INTERVENTIONS:
Drug: Indocyanine green for injection — ICG will be injected to participants preoperatively for molecular fluorescence image
  Other Names: ICG

SUMMARY:
The of this study is to explore the clinical outcomes of indocyanine green molecular fluorescence imaging in local resection of primary hepatocellular carcinoma (CNLC Ⅰa stage).

DETAILED DESCRIPTION:
Indocyanine green molecular imaging technique is often used in the surgical treatment of primary liver cancer. Its application in hepatectomy of primary liver cancer is currently in the stage of case accumulation and clinical research. No prospective study has been conducted to determine the clinical efficacy of indocyanine green molecular imaging for local hepatectomy of primary liver cancer. On the basis of more than 1000 liver resection procedures, the investigators want to apply indocyanine green molecular imaging technology, a cheap, simple and radiation-free method, to guide surgical resection. The purpose is to assist surgical procedures and improve participants' tumor-free survival.

ELIGIBILITY:
Inclusion Criteria:

* First clinical diagnosis of primary liver cancer (China liver cancer staging, CNLC Ia stage);
* Child-Pugh grading standard of liver function was GRADE A or B;
* 18-66 years old;
* Complete clinical case data;
* limited surgical methods (local resection);
* Voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

* There are basic diseases that cannot tolerate surgery (such as severe cardiopulmonary cerebral renal insufficiency);
* Tumor thrombus or distant metastasis was found in main portal vein and primary branch, main hepatic vein and branch, main hepatic vein and inferior vena cava by preoperative imaging examination;
* planned pregnancy, unplanned pregnancy and pregnancy;
* Preoperative child-Pugh grading standard of liver function was Grade C.
* Disease researchers that the investigator considers inappropriate to participate in this clinical trial.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
  No tumor recurrence within 3 years after surgery divided by total number of patients

SECONDARY OUTCOMES:
Positive margin rate | 14 days
  Compare positive margin rate in both groups
Negative margin rate | 14 days
  Compare negative margin rate in both groups
Length of the shortest cutting edge | 14 days
  The shortest distance between tumor and resection margin was compared between the two groups by pathological diagnosis
Operation time | 1 day
  Compare operation time in both groups
Intraoperative blood loss | 1 day
  Compare intraoperative blood loss in both groups
Intraoperative blood transfusion volume | 1 day
  Compare intraoperative blood transfusion volume in both groups
The number of small lesions of HCC | 14 days
  Small lesions detected by ICG fluorescence and confirmed by pathology in the intervention group
Residual tumor at the margin of liver cross-section | 14 days
  The number of residual tumors confirmed by ICG fluorescence detection at the liver margin of the intervention group
Intraoperative biliary fistula detection rate | 1 day
  The number of cases of successful intraoperative detection of biliary fistula by fluorescence in the intervention group divided by the total number of cases in the intervention group.
Extrahepatic metastases of primary hepatocellular carcinoma | 14 days
  The number of extrahepatic metastases of primary liver cancer detected by ICG and confirmed by pathology in the intervention group
Postoperative hospital stay | 30 days
  Compare Postoperative hospital stay in both groups. Eg: Postoperative hospital stay is the number of days from the day of surgery to the day of discharge.
Postoperative liver function index 1 | 5 days
  Compare the levels of Alanine aminotransferase on postoperative days 1, 3, and 5 in both groups
Postoperative liver function index 2 | 5 days
  Compare the levels of Aspartate aminotransferase on postoperative days 1, 3, and 5 in both groups
Postoperative liver function index 3 | 5 days
  Compare the levels of serum albumin on postoperative days 1, 3, and 5 in both groups
Postoperative liver function index 4 | 5 days
  Compare the levels of total bilirubin on postoperative days 1, 3, and 5 in both groups
Postoperative hemoglobin | 5 days
  Compare hemoglobin on postoperative days 1, 3, and 5 in both groups
Postoperative platelets | 5 days
  Compare platelets on postoperative days 1, 3, and 5 in both groups
Prothrombin time | 5 days
  Compare prothrombin time on postoperative days 1, 3, and 5 in both groups
Mortality rates | 3 months
  Perioperative death was defined as death occurring within 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chihua Fang, MD, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No